CLINICAL TRIAL: NCT00037895
Title: Stroke Rehabilitation Outcomes With Supported Treadmill Ambulation Training
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2340R
Record Dates: First submitted 2002-05-24; First posted 2002-05-27 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2002-05

CONDITIONS: Cerebrovascular Accident
Keywords: Stroke; Ambulation Training; Rehabilitation; Treadmill
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Procedure: Ambulation training

SUMMARY:
This project seeks to overcome the reduced walking capability, poor health status, decreased functional capacity, and sedentary lifestyle of stroke patients. The specific objectives are to compare the effects of regular inpatient stroke rehabilitation to regular rehabilitation combined with STAT after an acute stroke on: a) gait performance; b) functional outcomes; c) oxygen consumption during a seated task; and finally: d) using Brain Motor Control Assessment to obtain neurophysiological characteristics, as possible predictors of rehabilitation outcomes.

DETAILED DESCRIPTION:
Gait training is often delayed during the rehabilitation process because gait is thought to require preparation such as improved strength, balance, and coordination before the initiation of this more complex and demanding activity. We propose a new approach to perform early gait training with acute stroke patients, which consists of Supported Treadmill Ambulation Training (STAT) combined with conventional rehabilitation for achieving functional ambulation.

Hypotheses: This study will test three hypotheses;

1. The STAT group will develop greater gait speed, longer walking endurance, and lower oxygen costs for walking as compared to stroke patients receiving regular rehabilitation care.
2. The STAT group will develop better functional outcomes (Functional Independence Measurement total scores and on the transfers and locomotion subscales) as compared to stroke patients receiving regular rehabilitation care.
3. The STAT group will develop higher submaximal oxygen consumption as measured on a bicycle ergometer test compared to stroke patients receiving regular rehabilitation care.

Specific Objectives and Projected Timetable:

Since stroke patients have reduced walking capability, poor health status, decreased functional capacity, as well as a sedentary lifestyle, the specific objectives of this project are:

1. Compare the effects of regular inpatient stroke rehabilitation to regular stroke rehabilitation combined with STAT after an acute stroke on gait performance;
2. Compare the effects of regular inpatient stroke rehabilitation to regular rehabilitation combined with STAT after an acute stroke on functional outcomes, as defined by the Functional Independence Measure (FIM);
3. Compare the effects of regular inpatient stroke rehabilitation to regular stroke rehabilitation combined with STAT after an acute stroke on the oxygen consumption during a seated exercise task.
4. Explore whether neurophysiological characteristics using the Brain Motor Control Assessment (BMCA) predict rehabilitation outcomes.

Timetable: This 3-year project will compare the outcomes between two strategies of intervention during stroke rehabilitation. Admission, randomization, testing, intervention, reevaluation, and discharge will follow the time frame established by the facility while providing regular rehabilitation care for stroke patients. On average, the stroke rehabilitation process lasts two to three weeks.

ELIGIBILITY:
Recent unilateral stroke patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2001-01; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wolff, Ph.D., Special Assistant to the Director — Program Analysis and Review Section (PARS) VA Rehabilitation Research & Development Service; Danielle Kerkovitch, Ph.D. — Program Analysis and Review Section (PARS), VA Rehabilitation Research and development Service
Locations (1):
- VAMC, Houston, Texas, United States